CLINICAL TRIAL: NCT05435989
Title: Extended High-frequency Hearing and Speech Perception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Monson (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Brian Monson, Assistant Professor, University of Illinois at Urbana-Champaign
Organization: University of Illinois at Urbana-Champaign (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AH181; R01DC019745 (NIH)
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Low-pass Filtering Speech

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal-hearing listeners (Experimental)
  Interventions: Diagnostic Test: Reduced extended high-frequency audibility

INTERVENTIONS:
Diagnostic Test: Reduced extended high-frequency audibility — This study examines the effects of low-pass filtering speech on speech perception.

SUMMARY:
This study examines the effects of low-pass filtering speech on speech perception.

ELIGIBILITY:
Inclusion Criteria:

* native speakers of American English
* normal hearing 250-8000 Hz

Exclusion Criteria:

* non-native speakers of American English
* hearing loss

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Speech recognition or localization score | Day 1
  Speech recognition or localization scores are assessed using alternative forced choice procedures implemented with custom software scripts (e.g. in Matlab)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided